CLINICAL TRIAL: NCT00143910
Title: Measurement of Compliance in Renal Transplant Recipients
Brief Title: Natural History Study of Azathioprine Adherence
Status: Completed | Type: Observational
Sponsor: Thomas E. Nivens, MD (Individual)
Responsible Party: Sponsor
Organization: University of Minnesota (Other)
Other Study IDs: 9109M04306; NIH - DK13083
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Kidney Transplant
Keywords: Medication adherence; Patient compliance; Kidney transplant; Organ rejection; Allograft loss; Drug monitoring
MeSH Terms: conditions — Medication Adherence; Patient Compliance | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal transplant recipient: Recipients of successful renal transplant
  Interventions: Other: observation

INTERVENTIONS:
Other: observation

SUMMARY:
This study began in 1993 as a prospective, natural history study of renal transplant patients' medication compliance measured by using an electronic monitor on the cap of medication vials. Hypothesis: Poor medication compliance predicts adverse outcomes. Enrollment is closed.

DETAILED DESCRIPTION:
* The study is complete. Patient recruitment is closed and active patient involvement in the study has ended.
* Statistical analysis of monitor records and new patient outcome data continues

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient
* Discharged from hospital with functioning graft,not on dialysis
* Prescribed azathioprine

Exclusion Criteria:

* Unable to give informed consent
* Non English speaking
* Previous or concurrent organ transplant other than kidney
* Taking liquid form of azathioprine
* Followed outside of the United states

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Successful renal transplant recipients, discharged from hospital with a functioning renal transplant.
Sampling Method: Non-Probability Sample
Enrollment: 180
Dates: Start 1993-04; Primary Completion 1999-10 (Actual); Study Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
acute transplant rejection | 10 years

SECONDARY OUTCOMES:
Allograft loss | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Nevins, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Nevins TE, Kruse L, Skeans MA, Thomas W. The natural history of azathioprine compliance after renal transplantation. Kidney Int. 2001 Oct;60(4):1565-70. doi: 10.1046/j.1523-1755.2001.00961.x. PMID 11576374